CLINICAL TRIAL: NCT04037137
Title: Turkish Version of Caregiver Difficulties Scale: a Study of Reliability and Validity
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adıgüzel, Msc PhD. cd. Lecturer, Sanko University
Other Study IDs: Sanko M
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; Caregiver Burnout
Keywords: Caregiver Diffuculties Scale; reliability; validity; Turkish version
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Caregiver Difficulties Scale, Impact on Family Scale, WHOQOL-BREF Quality of Life Assessment, Nottingham Health Profile, Fatigue Severity Scale, Beck Depression Scale
  Other Names: assesment

SUMMARY:
As the life expectancy of individuals with Cerebral Palsy(CP) increases, their families' material, spiritual, physical and social difficulties increase, and in time, psychological and behavioral barriers occur in family members. While these barriers are increasing in developing countries, the whole family may be more vulnerable to the negative consequences of caring because of the limited availability of basic facilities for disabled people and the lack of temporary care services. The main aim of rehabilitation of individuals with CP is to improve their adaptive functions by increasing their postural control, locomotion and manipulative skills. Today, family-centered approaches for CP are known to be the most successful in terms of rehabilitation. Because the family is known to be of great importance in terms of active participation of the child in life. Therefore, while interdisciplinary treatments are in progress for the treatment of individuals, the success of rehabilitation is provided by interacting with the family, identifying their needs and problems and supporting them. There are many questionnaires developed to assess the difficulties experienced by the parents of individuals with CP. Of these, surveys adapted to Turkish are less common. The direct translation of the questionnaires into other languages does not guarantee its validity. If measures are to be used across cultures, it is known that the elements should not only be well translated linguistically, but also culturally adapted to maintain the content validity of the instrument across different cultures.

DETAILED DESCRIPTION:
Cerebral Palsy(CP) is a lifelong disability and 65-90% of these individuals have a normal lifespan. A multidisciplinary team approach is needed to evaluate and treat individuals with CP. This team varies according to the age, developmental level, severity of functional independence and participation in the society. However, according to the needs and dependency levels of individuals as well as team members, the family is at the center of the lives of these teams and their children. Depending on the limitations of their physical abilities, individuals with CP may need help from others in daily living activities (toilet, bath, mobilization, eating), although their limitations vary according to their clinical types. Therefore, CP can affect the lives of all family members. Today, it is known that especially the parents of individuals with CP experience widespread anxiety, financial problems, time-related pressures, and social-cultural activities. While some families adapt well, others may have difficulty coping and making various adjustments. This results in parents' life satisfaction, poor quality and deterioration of personal well-being. As a result of a study examining the quality of life; the importance of evaluating caregivers with reduced quality of life, potentially having physical, psychological or social problems. One of the effective ways of coping with the disabilities of a child with CP is to consider primary caregivers, especially mothers. Therefore, assessment of caregivers' responsibilities and their impact on health is a fundamental requirement of long-term care programs for children with disabilities. Paying special attention to caregivers can be achieved by using specific tools that determine their needs and, together with all family members, not only improve the quality of life of the child, but also accelerate the treatment of the child (9). It is necessary to assess the responsibilities of care in order to provide access to the necessary facilities by providing good support to the caregivers. This can only be achieved by having an appropriate scale of caregiver responsibilities (9). The use of questionnaires to assess caregivers is most common in developed countries. When the literature is examined, the scale called 'Caregiver Difficulties Scale (CDS) en which evaluates the responsibilities of the caregivers of the individuals with CP and covers the responsibilities in every aspect (10). A Turkish validity and reliability study of several questionnaires evaluating children with CP was conducted in Turkey (11). However, there is only one scale for Turkish validity and reliability studies on parental involvement (11). The aim of this study is to determine whether the Caregiver Difficulties Scale (CDS) is a valid and reliable tool by cultural adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Parents of individuals with CP receiving active treatment in a Special Education and Rehabilitation Center reported from Guidance and Research Centers after being diagnosed from all 2 nd and 3 rd health institutions in Gaziantep
* be willing to participate in the study

Exclusion Criteria:

* Having any diagnosed psychological disorder

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of individuals with CP patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Change of Caregiver Diffuculties Scale (CDS) | first day and 2 weeks later
  CDS is a self-administered questionnaire designed to be completed by the principal caregiver of the child with Cerebral palsy.The 4 subscales of CDS and the corresponding items are as follows.Concerns for the child, Impact on self, Support for caregiving, Support for caregiving.There is no definite cut off threshold for CDS; the total CDS score can be used to get an idea about the level of burden experienced by the caregivers, a higher score indicating a higher level of burden.CDS shows that a high CDS score (above 42) is predictive of caregiver psychological problems. Therefore, CDS is also useful as a potential screening tool for identification of caregivers who are at risk of psychological problems such as stress, depression and anxiety.After the second application,the consistency and problems of the CDS questionnaire were reviewed.
Impact on family scale | First day
  The original objective of the Impact on Family Scale is to assess the effect of a child's illness or health condition on the family. All items had astandard four-point scale ranging from strongly agree to strongly disagree.The four factors measured General Negative Impact (11 items), Disruption of Social Relations (nine items), Coping (four items), and Financial Impact (three items).Items are scored on a Likert scale.A low score indicates a higher impact of the chronic disease on the parents. Scores are calculated as percentages according to the highest scores of each part, using inverse proportion computing.

SECONDARY OUTCOMES:
Nottingham Health Profile | first day
  The NHP is an instrument designed to measure subjective health status containing 38items(answered "yes" or "no") that assess subjective distress in six subgroups:physical mobility (eight items), pain (eight items), sleep (five items), emotional reactions (nine items), social isolation (five items),and energy (three items). Scores for each subgroup range from 0 (no problem) to 100 (all problems listed were present).
Fatigue Severity Scale | first day
  The FSS, which was published in 1989 by Krupp, has nine items. For each question, the patient is asked to choose a number from 1 to 7 that indicates how much the patient agrees with each statement, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 4 or higher generally indicates severe fatigue.
Beck Depression Scale | first day
  This inventory comprises 21 questions, each with four possible answers (score: 0-3). If a symptom is more severe, the score will be higher. The higher the total score, the more depressed the patient.er the total score, the more depressed the patient. The Beck scores are divided in six grades of depression, according to the original description of the scores: 0-9: no or minimal depression 10-14: on the border of a depression 15-20: mild depression.21-30: mild-moderate depression. 31-40: moderate-severe depression. 41-63: severe depression.
WHOQOL-BREF quality of life assessment | first day
  WHOQOL-BREF was scored over four domains: Physical Capacity (7 items), Psychological Well-being (6 items), Social Relationship (4 items), and Environment (9 items). All items were rated on a 5-point scale with a higher score indicating a higher quality of life.Domain scores were calculated by multiplying the mean of all facet scores included in each domain by a factor of 4, and accordingly, potential scores for each domain ranged from 4-20.Responses from the two items of the Overall Quality of Life and General Health facet were calculated as a single score with a range of 4-20, as with the scoring method for the four domain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Adıgüzel, PhD cd., Principal Investigator — Sanko University; İpek Katırcı Kirmaci, PhD cd., Principal Investigator — Sanko University; Nevin Ergun, Prof., Principal Investigator — Sanko University; Suat Erel, Prof., Principal Investigator — Pamukkale University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)